CLINICAL TRIAL: NCT00066924
Title: Spirituality, Religiosity, and Immune Functioning
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Other Study IDs: F31AT001769-01 (NIH)
Record Dates: First submitted 2003-08-07; First posted 2003-08-08 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-05

CONDITIONS: Cancer; Depression; Dying Process
Keywords: spirituality; religiosity; immune functioning; psychoneuroimmunology; cytokines; cancer; death; depression
MeSH Terms: conditions — Neoplasms; Depression; Death

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to determine whether religiosity and spirituality are related to immune functioning, as measured by interleukin-6 blood plasma level, among terminally ill cancer patients.

ELIGIBILITY:
Inclusion criteria:

* Inpatient at Calvary Hospital
* Diagnosis of terminal cancer
* Score of 20 or above on Mini-Mental State Exam

Exclusion criteria:

* Presence of a psychiatric disorder that would preclude the production of meaningful data

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-09; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Barry Rosenfeld, PhD, Principal Investigator — Fordham University; William Breitbart, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Calvary Hospital, The Bronx, New York, United States

REFERENCES:
- [Background] McClain CS, Rosenfeld B, Breitbart W. Effect of spiritual well-being on end-of-life despair in terminally-ill cancer patients. Lancet. 2003 May 10;361(9369):1603-7. doi: 10.1016/S0140-6736(03)13310-7. PMID 12747880